CLINICAL TRIAL: NCT05336799
Title: Prevalence and Environmental Factors for Myopia Among Chinese School-aged Children and Adolescent in Tianjin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Tianjin Myopia Study
Record Dates: First submitted 2022-04-08; First posted 2022-04-20 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Myopia; Refractive Errors
Keywords: Myopia; Socioeconomics
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The high prevalence of myopia has become a global public health problem. The study amied to investigate the prevalence and progression of myopia associated with social environmental factors in Tianjin, a Chinese megacity in north China.

DETAILED DESCRIPTION:
The high prevalence of myopia has become a global public health problem, especially in East and South Asian countries. It's still not clear for the prevalence and progression of myopia associated with social environmental factors. Thus, the investigators will conducted a long-term observational study to the effect of the socioeconomics, medical resources and school-related environmental parameters and others on the prevalence and progression of myopia among Chinese school-aged children and adolescent.

ELIGIBILITY:
Inclusion Criteria:

* aged 6 to 18 years
* no ocular diseases and systemic diseases
* consent to undergo an eye examination

Exclusion Criteria:

* schoolchildren unwilling to participate

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All school-aged children and adolescents completed the vision screening in the included school.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of myopia | up to 3years
  Myopia is defined as any eye's SER (sphere + 1/2 cylinder) of at least -0.5 diopters (D).

SECONDARY OUTCOMES:
Changes in prevalence of myopia | up to 3years
  Myopia is defined as any eye's SER (sphere + 1/2 cylinder) of at least -0.5 diopters (D).
Changes of Spherical equivalent | changes from baseline at 36months
  Changes of Spherical equivalent

CONTACTS AND LOCATIONS:
Overall Officials: yan wang, Study Chair — Tianjin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morgan IG, French AN, Ashby RS, Guo X, Ding X, He M, Rose KA. The epidemics of myopia: Aetiology and prevention. Prog Retin Eye Res. 2018 Jan;62:134-149. doi: 10.1016/j.preteyeres.2017.09.004. Epub 2017 Sep 23. PMID 28951126
- [Background] Guo Y, Liu LJ, Xu L, Lv YY, Tang P, Feng Y, Meng M, Jonas JB. Outdoor activity and myopia among primary students in rural and urban regions of Beijing. Ophthalmology. 2013 Feb;120(2):277-83. doi: 10.1016/j.ophtha.2012.07.086. Epub 2012 Oct 23. PMID 23098368
- [Background] Tenovuo J, Mielityinen H, Paunio K. The effect of dental plaque grown in the presence of xylitol or sucrose on bone resorption in vitro. Pharmacol Ther Dent. 1981;6(1-2):35-43. PMID 6941318